CLINICAL TRIAL: NCT05814705
Title: Comparison of High-protein Formulation With/Without Urolithin a During a Unilateral Knee Immobilization: a Pilot Proof-of-concept Trial
Brief Title: The Effects of Protein Supplementation With or Without Urolithin A During Single-leg Immobilization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13783; ISRCTN20052152 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2023-03-10; First posted 2023-04-18 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Healthy; Muscle Disuse Atrophy
MeSH Terms: conditions — Muscular Disorders, Atrophic | interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein supplement (Active Comparator)
  Interventions: Dietary Supplement: Protein supplement
- Protein supplement with Urolithin A (Experimental)
  Interventions: Dietary Supplement: Protein supplement with Urolithin A

INTERVENTIONS:
Dietary Supplement: Protein supplement — Ready-to-drink protein beverage consumed once daily for 28 days
  Arms: Protein supplement
Dietary Supplement: Protein supplement with Urolithin A — Ready-to-drink protein beverage with 1000 mg of Urolithin A consumed once daily for 28 days
  Arms: Protein supplement with Urolithin A

SUMMARY:
There are times in life when people cannot use their muscles, such as during illness or injury. Muscle and mitochondria (the 'energy factory' in cells) health decline very quickly when people cannot use their muscles, but certain foods can help reduce these declines. Recent research suggests that Urolithin A, which is a natural compound that can be produced after eating pomegranates, nuts, and berries, improves muscle health. In this study, the investigators aim to investigate if a protein beverage (standard care during disuse) with or without Urolithin A can reduce or prevent the loss of muscle health while wearing a knee brace (muscle disuse).

DETAILED DESCRIPTION:
After participants provide informed consent to participate and are deemed eligible for the study (Day 0), participants will sequentially complete the three phases of this study:

1. RUN-IN phase: participants continue habitual lifestyle (Day 7-Day 14 [1 week])
2. IMMOBILIZATION phase: participants undergo 2 weeks of unilateral knee immobilization (Day 14-Day 28 [2 weeks])
3. RECOVERY phase: participants return to habitual lifestyle (Day 28-Day 35 [1 week])

Participants will consume their randomly assigned supplement daily during all three phases.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18-30 years
2. Healthy, non-smoking
3. BMI between 20 and 30 kg/m^2
4. No orthopedic issues that would preclude participation in the knee bracing protocol
5. Not taking any medication or with any medical condition that, in the opinion of the investigators, would compromise the study outcome or the safety of the research participant
6. Provide informed consent
7. Understand COVID-19 risks and procedures for in person research and sign Information Letter: COVID-19 Risks and Procedures for In-Person Research at McMaster University

Exclusion Criteria:

1. Subject has any concurrent medical, orthopedic, or psychiatric requirements that, in the opinion of the investigators, would compromise their ability to comply with the study requirements
2. Clinically significant abnormal laboratory results at screening
3. Participation in a clinical research trial within 30 days before randomization
4. Allergy or sensitivity to study ingredients
5. Individuals who are cognitively impaired and/or who are unable to give informed consent
6. Any other condition that, in the opinion of the investigators, may adversely affect the subject's ability to complete the study or its measures or may pose a significant risk to the subject
7. Any cachexia-related condition or any genetic muscle diseases or disorders
8. Current gastrointestinal condition that could interfere with the study (e.g., IBS/IBD [irritable bowel syndrome/inflammatory bowel disease], diarrhea, acid reflux disease, dysphagia, etc.)
9. Excessive alcohol consumption (>21 units/week) and/or a smoker (cigarettes or vaping)
10. Concomitant use of corticosteroids, antibiotics, any anabolic steroid, creatine, whey protein supplements, casein, branched-chain amino acids (BCAAs) or any other NHP [Natural Health Product], medication or supplement used for muscle strengthening/building within 45 days prior to screening
11. Contraindications to an MRI scan (metal implants, metal-based ink tattoo)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in maximal mitochondrial respiration (rate of oxygen flux) and mitochondrial ADP [adenosine diphosphate] sensitivity (Oroboros O2k) | Outcome measured and reported for: Day 7, Day 14, Day 28, Day 35
  Oxygen flux in muscle measured using Oroboros

SECONDARY OUTCOMES:
Muscle strength (Biodex) | Day 7, Day 14, Day 28, Day 35
  Isometric leg extension strength
Quadriceps muscle size | Outcome measured and reported for: Day 14, Day 28, Day 35
  Muscle size measured using MRI
Muscle protein fractional synthetic rate | Day 7, Day 14, Day 28, Day 35; integrated synthesis rates reported for Day 7-14, Day 14-28; Day 28-35
  Protein synthetic rate using labelled alanine incorporation

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No